CLINICAL TRIAL: NCT02512302
Title: A Crossover Clinical Pharmacology Study to Evaluate the Total Systemic Exposure and Lung Bioavailability of SUN-101 and Seebri® Breezhaler® Administered With and Without Activated Charcoal in Subjects With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Study to Determine the Amount of Glycopyrrolate Absorbed in the Lungs After Taking the Medicine With a eFlow Nebulizer and Seebri® Breezhaler® With and Without Activated Charcoal in Subjects With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD).
Acronym: GOLDEN7
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunovion Respiratory Development Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SUN101-105
Record Dates: First submitted 2015-07-24; First posted 2015-07-30 (Estimated); Results first posted 2018-09-14 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-09

CONDITIONS: COPD
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Glycopyrrolate; Charcoal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- SUN-101 via eFlow nebulizer (Experimental): 50 mcg glycopyrrolate via Electronic Nebulizer
  Interventions: Drug: SUN-101 via eFlow nebulizer
- SUN-101 via eFlow nebulizer with activated charcoal (Experimental): 50 mcg glycopyrrolate via Electronic Nebulizer with activated charcoal
  Interventions: Drug: SUN-101 via eFlow nebulizer with activated charcoal
- Seebri® Breezhaler® (Active Comparator): 63 mcg glycopyrronium bromide (50 mcg glycopyrronium) via DPI
  Interventions: Drug: Seebri® Breezhaler®
- Seebri® Breezhaler® with activated charcoal (Active Comparator): : : 63 mcg glycopyrronium bromide (50 mcg glycopyrronium) via DPI with activated charcoal
  Interventions: Drug: Seebri® Breezhaler® with activated charcoal
- : Glycopyrrolate Injection (Active Comparator): 50 mcg glycopyrrolate via IV infusion
  Interventions: Drug: Glycopyrrolate Injection

INTERVENTIONS:
Drug: SUN-101 via eFlow nebulizer — 50 mcg glycopyrrolate via Electronic Nebulizer
  Other Names: Glycopyrrolate
  Arms: SUN-101 via eFlow nebulizer
Drug: SUN-101 via eFlow nebulizer with activated charcoal — 50 mcg glycopyrrolate via Electronic Nebulizer with activated charcoal
  Other Names: Glycopyrrolate
  Arms: SUN-101 via eFlow nebulizer with activated charcoal
Drug: Seebri® Breezhaler® — 63 mcg glycopyrronium bromide (50 mcg glycopyrronium) via DPI
  Other Names: glycopyrronium, glycopyrronium bromide
  Arms: Seebri® Breezhaler®
Drug: Seebri® Breezhaler® with activated charcoal — 63 mcg glycopyrronium bromide (50 mcg glycopyrronium) via DPI with activated charcoal
  Other Names: glycopyrronium, glycopyrronium bromide
  Arms: Seebri® Breezhaler® with activated charcoal
Drug: Glycopyrrolate Injection — 50 mcg glycopyrrolate via IV
  Other Names: Glycopyrrolate
  Arms: : Glycopyrrolate Injection

SUMMARY:
The purpose of this research study is to determine the amount of medicine absorbed in the lungs following dosing via eFlow nebulizer and Seebri® Breezhaler® with and without activated charcoal in subjects with moderate to severe chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
This is a randomized, open-label, single-dose per dosing period, five-way crossover study in subjects 40 to 70 years of age with a diagnosis of moderate to severe COPD per Global Initiative for Chronic Obstructive Lung Disease guidelines. After a subject provides consent for study participation, there will be a Screening Period lasting up to 3 weeks to determine study eligibility and to allow for appropriate washout of prohibited medications.

Eligible subjects will be randomized to one of 10 treatment Sequences. There will be a minimum of a 7-day washout period between each treatment visit. At each visit, subjects will receive one dose of study medication according to the sequence assigned.

Subjects with a ≥ 20% decrease in forced expiratory volume in one second (FEV1) based on review of the Visit predose value compared with the Screening value will be evaluated by the investigator for continuation in the study.

Subjects taking theophylline will not be able to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 40 to 70 years-old, inclusive.
2. A clinical diagnosis of moderate to severe COPD according to the GOLD 2014 guidelines.
3. Current smokers or ex-smokers with at least 10 pack-year smoking history (eg, at least 1 pack/day for 10 years, or equivalent).
4. Post-bronchodilator (following inhalation of ipratropium bromide) FEV1 ≥ 30% and ≤ 80% of predicted normal during the Screening Period.
5. Post-bronchodilator (following inhalation of ipratropium bromide) FEV1/FVC ratio ≤ 0.70 during the Screening Period.
6. Ability to perform reproducible spirometry according to the American Thoracic Society (ATS) and/or European Respiratory Society (ERS) guidelines (2005).
7. Subject, if female ≤ 70 years of age and of child bearing potential, must have a negative urine pregnancy test at Visit 1. Females of childbearing potential must be instructed to and agree to avoid pregnancy during the study and must use an acceptable method of birth control: a) an oral contraceptive, an intrauterine device (IUD), implantable contraceptive, transdermal or injectable contraceptive for at least 1 month prior to entering the study with continued use throughout the study and for thirty days following participation; b) barrier method of contraception, eg, condom and /or diaphragm with spermicide while participating in the study; and/or c) abstinence.
8. Willing and able to remain at the study site for at least 24 hours for each treatment day.
9. Willing and able to provide written informed consent.
10. Willing and able to attend all study visits and adhere to all study assessments and procedures.

Exclusion Criteria:

1. Severe comorbidities including unstable cardiac or pulmonary disease or any other medical conditions that would, in the opinion of the Investigator, preclude the subject from safely completing the required tests or the study, or is likely to result in disease progression that would require withdrawal of the subject, included but not limited to the following:

   * Unstable ischemic heart disease (diagnosis of myocardial infarction or admission for acute coronary syndrome) within 6 months of screening.
   * Unstable cardiac arrhythmia or heart failure (change in treatment plan) within 6 months.
   * Treatment for diabetes mellitus within 6 months of screening.
2. Current evidence or history of a clinically significant abnormality of cardiac rhythm and/or conduction findings.
3. Concomitant clinically significant respiratory disease other than COPD (eg, asthma, tuberculosis, bronchiectasis, or other non-specific pulmonary disease).
4. History of malignancy of any organ system treated or untreated within the past 5 years, with the exception of localized basal cell carcinoma of the skin.
5. Recent history of COPD exacerbation requiring hospitalization or need for increased treatments for COPD within 6 weeks prior to the Screening Period.
6. Use of daily oxygen therapy > 10 hours per day.
7. Use of oral, intravenous, or intramuscular steroids within 3 months prior to the Screening Period.
8. Respiratory tract infection within 6 weeks prior to or during the Screening Period.
9. Significant blood loss (> 500 mL) or donated blood within 60 days preceding screening or plans to donate blood within 60 days after completing the study.
10. History of or clinically significant ongoing bladder outflow obstruction or history of catheterization for relief of bladder outflow obstruction within the previous 6 months.
11. History of narrow-angle glaucoma.
12. Prolonged QTc interval (> 450 msec for males and > 470 msec for females) during the Screening Period, or history of long QT syndrome.
13. Recent documented history (previous 12 months) of substance abuse.
14. .Positive urine drug screen at Visit 1 provided the subject is unable to produce a valid medical rationale for the test result (eg, prescription medication).
15. Positive HbsAg, Hepatitis C antibody, or HIV 1/2 antibody test at Screening.
16. History of hypersensitivity or intolerance to aerosol medications, β2-agonists, anticholinergics, or sympathomimetic amines.
17. Significant psychiatric disease that would likely result in the subject not being able to complete the study, in the opinion of the Investigator.
18. Participation in another investigational drug study where drug was received within 30 days prior to the Screening Period, or current participation in another investigational drug trial in which study treatment is being administered, including a SUN-101 study
19. Previously received SUN-101 (active treatment; formerly known as EP-101).
20. Previously received any glycopyrrolate product within 28 days of Screening.
21. Subject is taking theophylline.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Head of Global Clinical, Respiratory and Bio-threapeutics, Study Chair — Sunovion Pharmaceuticals
Locations (2):
- United Kingdom (2):
  - Queen Anne Street Medical Center, London
  - Medicines evaluation Unit Ltd., Manchester

REFERENCES:
- [Derived] Leaker BR, Singh D, Nicholson GC, Hezelova B, Goodin T, Ozol-Godfrey A, Galluppi G, Barnes PJ. Evaluation of systemic absorption and bronchodilator effect of glycopyrronium bromide delivered by nebulizer or a dry powder inhaler in subjects with chronic obstructive pulmonary disease. Respir Res. 2019 Jun 28;20(1):132. doi: 10.1186/s12931-019-1113-z. PMID 31253162

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible subjects will be randomized to one of 10 treatment sequences. There will be a minimum of a 7-day washout period between each treatment visit. At each visit, subjects will receive one dose of study medication according to the sequence assigned.
Groups:
- Treatment Group One: Participants received Seebri Breezhaler with activated charcoal 63 mcg; SUN-101 50 mcg via eFlow nebulizer with activated charcoal; Glycopyrrolate injection via IV infusion; SUN-101 50 mcg via e flow nebulizer; Seebri Breezhaler 63 mcg for each of the five treatment periods
- Treatment Group Two: Participants received SUN-101 50 mcg via eFlow nebulizer, SUN-101 50 mcg via eFlow nebulier with activated charcoal; Seebri Breezhaler 63 mcg, Seebri Breezhaler 63 mcg with activated charcoal; Glycopyrrolate injection via IV infusion for each of the five treatment periods
- Treatment Group Three: Participants recveived SUN-101 50 mcg via eFlow nebulizer; Seebri Breezhaler 63mcg; SUN-101 50mcg via eFlow nebulizer with activated charcoal; Glycopyrrolate injection via IV infusion; Seebri Breezerhaler 63mcg with activated charcoal for each of the five treatment periods
- Treatment Group Four: Participants received Glycopyrrolate injection via IV infusion; Seebri Breezhaler 63mcg with activated charcoal; Seebri Breezhaler 63mcg; SUN-101 50 mcg via eFlow nebulizer with activated charcoal; SUN-101 50 mcg via eFlow nebulizer for each of the five treatment periods
- Treatment Group Five: Participants received Seebri Breezhaler 63mcg ; Glycopyrrolate injection via IV infusion; SUN-101 50 mcg via eFlow nebulizer; Seebri Breezhaler 63mcg with activated charcoal; SUN-101 50 mcg via eFlow nebulizer with activated charcoal; for each of the five treatment periods
- Treatment Group Six: Participants received Seebri Breezhaler 63mcg with activated charcoal ; Glycopyrrolate injection via IV infusion; SUN-101 50 mcg via eFlow nebulizer with activated charcoal; Seebri Breezhaler 63mcg SUN-101 50 mcg via eFlow nebulizer for each of the five treatment periods
- Treatment Group Seven: Participants received Seebri Breezhaler 63mcg ; SUN-101 50 mcg via eFlow nebulizer; Glycopyrrolate injection via IV infusion; SUN-101 50 mcg via eFlow nebulizer with activated charcoal; Seebri Breezhaler 63mcg with activated charcoal for each of the five treatment periods
- Treatment Group Eight: Participants received SUN-101 50 mcg via eFlow nebulizer with activated charcoal; SUN-101 50 mcg via eFlow nebulizer; Seebri Breezhaler 63mcg with activated charcoal; Seebri Breezhaler 63 mcg; Glycopyrrolate injection via IV infusion for each of the five treatment periods
- Treatment Group Nine: Participants received Glycopyrrolate injection via IV infusion; Seebri Breezhaler 63 mcg; Seebri Breezhaler 63mcg with activated charcoal; SUN-101 50 mcg via eFlow nebulizer SUN-101 50 mcg via eFlow nebulizer with activated charcoalfor each of the five treatment periods
- Treatment Group Ten: Participants received SUN-101 50 mcg via eFlow nebulizer with activated charcoal; Seebri Breezhaler 63mcg with activated charcoal; SUN-101 50 mcg via eFlow nebulizer; Glycopyrrolate injection via IV infusion;Seebri Breezhaler 63mcg for each of the five treatment periods
Period: Period 1
Arm/Group | Treatment Group One | Treatment Group Two | Treatment Group Three | Treatment Group Four | Treatment Group Five | Treatment Group Six | Treatment Group Seven | Treatment Group Eight | Treatment Group Nine | Treatment Group Ten
Started | 3 | 3 | 4 | 3 | 3 | 3 | 2 | 3 | 3 | 3
Completed | 3 | 2 | 4 | 3 | 3 | 3 | 2 | 3 | 3 | 3
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Treatment Group One | Treatment Group Two | Treatment Group Three | Treatment Group Four | Treatment Group Five | Treatment Group Six | Treatment Group Seven | Treatment Group Eight | Treatment Group Nine | Treatment Group Ten
Started | 3 | 2 | 4 | 3 | 3 | 3 | 2 | 3 | 3 | 3
Completed | 3 | 2 | 4 | 3 | 3 | 3 | 2 | 3 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Period 3
Arm/Group | Treatment Group One | Treatment Group Two | Treatment Group Three | Treatment Group Four | Treatment Group Five | Treatment Group Six | Treatment Group Seven | Treatment Group Eight | Treatment Group Nine | Treatment Group Ten
Started | 3 | 2 | 4 | 3 | 3 | 3 | 2 | 3 | 3 | 2
Completed | 3 | 2 | 3 | 3 | 3 | 3 | 2 | 3 | 3 | 2
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Treatment Group One | Treatment Group Two | Treatment Group Three | Treatment Group Four | Treatment Group Five | Treatment Group Six | Treatment Group Seven | Treatment Group Eight | Treatment Group Nine | Treatment Group Ten
Started | 3 | 2 | 3 | 3 | 3 | 3 | 2 | 3 | 3 | 2
Completed | 3 | 2 | 3 | 3 | 3 | 3 | 1 | 3 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Period 5
Arm/Group | Treatment Group One | Treatment Group Two | Treatment Group Three | Treatment Group Four | Treatment Group Five | Treatment Group Six | Treatment Group Seven | Treatment Group Eight | Treatment Group Nine | Treatment Group Ten
Started | 3 | 2 | 3 | 3 | 3 | 3 | 1 | 3 | 3 | 2
Completed | 3 | 2 | 3 | 3 | 3 | 3 | 1 | 3 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total number of participants from all treatment groups
Arm/Group | Total
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 28
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 30

OUTCOME MEASURES:

1. Primary Outcome: Cmax
Description: maximum observed concentration-Cmax is calculated from plasma concentrations analyzed from blood samples collected between 0 and 48 hr.
Time Frame: Up to Week 5
Population: The Pharmacokinetic (PK) population consists of all subjects who were randomized, received study medication and have any evaluable PK data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Pg/mL
Arm/Group | SUN-101 Via eFlow Nebulizer | SUN-101 Via eFlow Nebulizer With Activated Charcoal | Seebri® Breezhaler® | Seebri® Breezhaler® With Activated Charcoal | : Glycopyrrolate Injection
Number analyzed (Participants) | 29 | 29 | 28 | 26 | 27
Pg/mL | 53.75 (51.746) | 49.27 (60.996) | 166.79 (76.348) | 148.03 (39.841) | 3787.47 (115.166)

2. Primary Outcome: Area Under the Curve From Time Zero to 24 Hours (AUC0_24)
Description: Area under the drug concentration-time curve from time zero to 24 hours postdose pk parameteres are calculated from plasma concentration analyzed from blood samples collected between 0 and 48 hr
Time Frame: Up to Week 5
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*pg/mL
Arm/Group | SUN-101 Via eFlow Nebulizer | SUN-101 Via eFlow Nebulizer With Activated Charcoal | Seebri® Breezhaler® | Seebri® Breezhaler® With Activated Charcoal | : Glycopyrrolate Injection
Number analyzed (Participants) | 29 | 29 | 28 | 26 | 27
hr*pg/mL | 172.23 (100.974) | 159.12 (92.720) | 472.35 (90.233) | 428.52 (46.985) | 1961.79 (142.488)

3. Primary Outcome: Area Under the Curve From Time Zero to Infinity (AUC0_infinity)
Description: calculated by summing AUC0-last and the AUC extrapolated from tlast to infinity: AUC0-∞ = AUC0-last+ Clast / | λz | Clast / | λz | is the extrapolated area under the curve from tlast to infinity. If this quantity is greater than 20% of AUC0-∞, then AUC0-∞ was considered to be missing.
  Pk parameters are calculated from plasma concentration analyzed from blood samples collected between 0 and 48 hr.
Time Frame: Up to Week 5
Population: The Pharmacokinetic (PK) population consists of all subjects who were randomized, received study medication, and have any evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*pg/mL
Arm/Group | SUN-101 Via eFlow Nebulizer | SUN-101 Via eFlow Nebulizer With Activated Charcoal | Seebri® Breezhaler® | Seebri® Breezhaler® With Activated Charcoal | : Glycopyrrolate Injection
Number analyzed (Participants) | 8 | 6 | 15 | 10 | 21
hr*pg/mL | 234.23 (77.206) | 167.84 (41.208) | 607.53 (79.340) | 570.90 (63.913) | 2550.85 (117.068)

4. Secondary Outcome: Clearance (CL) for IV Infusion of 50 mcg of Glycopyrrolate
Description: calculated as Dose/AUC0-inf after the IV dose administration. If AUC0-inf is missing, then CL was considered as missing.
  Pk parameters are calculated from plasma concentration analyzed from blood samples collected between 0 and 48 hr.
Time Frame: Up to Week 5
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters/hr
Arm/Group | : Glycopyrrolate Injection
Number analyzed (Participants) | 21
Liters/hr | 19.60 (117.068)

5. Secondary Outcome: Volume of Distribution During the Elimination Phase (Vz) for IV Infusion of 50 mcg of Glycopyrrolate
Description: calculated as Dose/(AUC0-inf*λz). Pk parameters are calculated from plasma concentration analyzed from blood samples collected between 0 and 48 hr.
Time Frame: Up to Week 5
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | : Glycopyrrolate Injection
Number analyzed (Participants) | 21
Liters | 113.06 (131.141)

6. Secondary Outcome: Time of Occurrence of Cmax (Tmax) for IV Infusion of 50 mcg of Glycopyrrolate
Description: The time 0 is based on start of the infusion. Pk parameters are calculated from plasma concentration analyzed from blood samples collected between 0 and 48 hr.
Time Frame: Up to Week 5
Population: as for outcome 3
Measure: Median (Full Range); unit: hr
Arm/Group | : Glycopyrrolate Injection
Number analyzed (Participants) | 27
hr | 0.100 [0.08 to 0.40]

7. Secondary Outcome: Terminal Half Life (t1/2) for IV Infusion of 50 mcg of Glycopyrrolate
Description: calculated as ln(2) / λz . At least 3 data points at the terminal elimination phase were required to determine t½.
  Pk parameters are calculated from plasma concentration analyzed from blood samples collected between 0 and 48 hr.
Time Frame: Up to Week 5
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | : Glycopyrrolate Injection
Number analyzed (Participants) | 21
hr | 3.998 (111.8589)

8. Secondary Outcome: Area Under the Curve Zero to 48 Hours (AUC0_48) for Seebri Breezhaler and Sun-101 AUC0-48, CL/F, Vz/F, Tmax, t½, and Dose Normalized Cmax, AUC0-24, AUC0-48, AUC0-∞ - AUC0-∞ -
Description: Area under the drug concentration-time curve from time zero to 48 hours postdose Pk parameters are calculated from plasma concentration analyzed from blood samples collected between 0 and 48 hr.
Time Frame: Up to Week 5
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*pg/mL
Arm/Group | SUN-101 Via eFlow Nebulizer | SUN-101 Via eFlow Nebulizer With Activated Charcoal | Seebri® Breezhaler® | Seebri® Breezhaler® With Activated Charcoal
Number analyzed (Participants) | 29 | 29 | 28 | 26
hr*pg/mL | 182.59 (112.339) | 179.78 (108.906) | 524.18 (99.365) | 485.99 (56.588)

9. Secondary Outcome: Apparent Clearance Calculated as Dose/AUC0-INF After Extravascular Dose Administration of Seebri Breezhaler and SUN-101
Description: calculated as Dose/AUC0-∞ after extravascular dose administration, where F = Bioavailability. If AUC0-∞ is missing, then CL/F is considered as missing.
  Pk parameters are calculated from plasma concentration analyzed from blood samples collected between 0 and 48 hr.
Time Frame: up to week 5
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | SUN-101 Via eFlow Nebulizer | SUN-101 Via eFlow Nebulizer With Activated Charcoal | Seebri® Breezhaler® | Seebri® Breezhaler® With Activated Charcoal
Number analyzed (Participants) | 8 | 6 | 15 | 10
L/hr | 213.47 (77.206) | 297.91 (41.208) | 103.70 (79.340) | 110.35 (63.913)

10. Secondary Outcome: Apparent Volume of Distribution (Vz/F) After Extravascular Dose Administration of Seebri Breezhaler and SUN-101
Description: calculated as Dose/(AUC0-∞* λz), where F = Bioavailability. If AUC0-∞ is missing, then Vz/F is considered as missing.
  Pk parameters are calculated from plasma concentration analyzed from blood samples collected between 0 and 48 hr
Time Frame: up to week 5
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | SUN-101 Via eFlow Nebulizer | SUN-101 Via eFlow Nebulizer With Activated Charcoal | Seebri® Breezhaler® | Seebri® Breezhaler® With Activated Charcoal
Number analyzed (Participants) | 8 | 6 | 15 | 10
liters | 1263.63 (31.716) | 1668.59 (17.994) | 1305.30 (23.585) | 1708.81 (22.543)

11. Secondary Outcome: Time of Occurrence of Cmax (Tmax) for Seebri Breezhaler and SUN-101
Description: The time 0 is based on start of the inhalation. Pk parameters are calculated from plasma concentration analyzed from blood samples collected between 0 and 48 hr.
Time Frame: up to week 5
Population: as for outcome 3
Measure: Median (Full Range); unit: hr
Arm/Group | SUN-101 Via eFlow Nebulizer | SUN-101 Via eFlow Nebulizer With Activated Charcoal | Seebri® Breezhaler® | Seebri® Breezhaler® With Activated Charcoal
Number analyzed (Participants) | 29 | 29 | 28 | 26
hr | 0.317 [0.08 to 12.05] | 0.250 [0.07 to 12.3] | 0.250 [0.03 to 1.57] | 0.250 [0.05 to 0.40]

12. Secondary Outcome: Terminal Half Life (t1/2) for for Seebri Breezhaler and SUN-101
Description: as for outcome 7
Time Frame: up to week 5
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | SUN-101 Via eFlow Nebulizer | SUN-101 Via eFlow Nebulizer With Activated Charcoal | Seebri® Breezhaler® | Seebri® Breezhaler® With Activated Charcoal
Number analyzed (Participants) | 13 | 10 | 20 | 20
hr | 6.554 (135.6286) | 5.191 (61.4971) | 10.378 (80.1891) | 14.866 (69.3836)

13. Secondary Outcome: Dose Normalized Cmax for Seebri and SUN-101.
Description: Maximum observed concentration multiplied by the dose normalization factor. Pk parameters are calculated from plasma concentration analyzed from blood samples collected between 0 and 48 hr.
  The dose normalization factor calculation has two components: dose equivalent glycopyrrolate amount and the delivery efficiency (% dose delivered). For Sun-101 50 mcg, the dose normalization factor is 1.59, for Seebri Breezhaler it is 0.9.
Time Frame: up to week 5
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Pg/mL
Arm/Group | SUN-101 Via eFlow Nebulizer | SUN-101 Via eFlow Nebulizer With Activated Charcoal | Seebri® Breezhaler® | Seebri® Breezhaler® With Activated Charcoal
Number analyzed (Participants) | 29 | 29 | 28 | 26
Pg/mL | 85.46 (51.746) | 78.33 (60.996) | 150.11 (76.348) | 133.22 (39.841)

14. Secondary Outcome: Dose Normalized Area Under the Curve Zero to 24 Hours (AUC0_24) for Seebri and SUN-101
Description: Pk parameters are calculated from plasma concentration analyzed from blood samples collected between 0 and 48 hr.
  Area under the drug concentration-time curve from time zero to 24 hours postdose multiplied by the dose normalization factor. The dose normalization factor calculation has two components: dose equivalent glycopyrrolate amount and the delivery efficiency (% dose delivered). For Sun-101 50 mcg, the dose normalization factor is 1.59, for Seebri Breezhaler it is 0.9.
Time Frame: up to week 5
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*pg/mL
Arm/Group | SUN-101 Via eFlow Nebulizer | SUN-101 Via eFlow Nebulizer With Activated Charcoal | Seebri® Breezhaler® | Seebri® Breezhaler® With Activated Charcoal
Number analyzed (Participants) | 29 | 29 | 28 | 26
hr*pg/mL | 273.85 (100.974) | 253.00 (92.720) | 425.12 (90.233) | 385.67 (46.985)

15. Secondary Outcome: Dose Normalized Area Under the Curve Zero to 48 Hours (AUC0_48) for Seebri and SUN-101
Description: Pk parameters are calculated from plasma concentration analyzed from blood samples collected between 0 and 48 hr.
  Area under the drug concentration-time curve from time zero to 48 hours postdose multiplied by the dose normalization factor. The dose normalization factor calculation has two components: dose equivalent glycopyrrolate amount and the delivery efficiency (% dose delivered). For Sun-101 50 mcg, the dose normalization factor is 1.59, for Seebri Breezhaler it is 0.9.
Time Frame: up to week 5
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*pg/mL
Arm/Group | SUN-101 Via eFlow Nebulizer | SUN-101 Via eFlow Nebulizer With Activated Charcoal | Seebri® Breezhaler® | Seebri® Breezhaler® With Activated Charcoal
Number analyzed (Participants) | 29 | 29 | 28 | 26
hr*pg/mL | 290.32 (112.339) | 285.85 (108.906) | 471.76 (99.365) | 437.39 (56.588)

16. Secondary Outcome: Dose Normalized Area Under the Curve Zero From Zero to Infinity (AUC0_inf) for Seebri and SUN-101
Description: Pk parameters are calculated from plasma concentration analyzed from blood samples collected between 0 and 48 hr.
  Area under the drug concentration-time curve from zero to infinity, calculated by summing AUC0-last and the AUC extrapolated from tlast to infinity multiplied by the dose normalization factor: dose normalization factor* (AUC0-∞ = AUC0-last+ Clast / | λz | ) Clast / | λz | is the extrapolated area under the curve from tlast to infinity. If this quantity is greater than 20% of AUC0-∞, then AUC0-∞ was considered to be missing.
  The dose normalization factor calculation has two components: dose equivalent glycopyrrolate amount and the delivery efficiency (% dose delivered). For Sun-101 50mcg , the dose normalization factor is 1.59, for Seebri Breezhaler it is 0.9.
Time Frame: up to week 5
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*pg/mL
Arm/Group | SUN-101 Via eFlow Nebulizer | SUN-101 Via eFlow Nebulizer With Activated Charcoal | Seebri® Breezhaler® | Seebri® Breezhaler® With Activated Charcoal
Number analyzed (Participants) | 8 | 6 | 15 | 10
hr*pg/mL | 372.42 (77.206) | 266.86 (41.208) | 546.78 (79.340) | 513.81 (63.931)

17. Secondary Outcome: The Number of Subjects With Adverse Events (AEs), Serious Adverse Events (SAEs), and AEs Leading to Discontinuation
Description: An adverse event (AE) that occurred on or after the first dose of study medication, any AE with a missing start date and a stop date on or after the first dose of study medication, or any AE with both a missing start and stop date.
Time Frame: Up to Week 5
Population: Safety population was defined as all subjects who were randomized to treatment and received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | SUN-101 Via eFlow Nebulizer | SUN-101 Via eFlow Nebulizer With Activated Charcoal | Seebri® Breezhaler® | Seebri® Breezhaler® With Activated Charcoal | : Glycopyrrolate Injection
Number analyzed (Participants) | 29 | 29 | 28 | 27 | 27
participants
  Adverse Events | 6 | 9 | 7 | 11 | 7
  Serious Adverse Events | 0 | 0 | 0 | 0 | 0
  Adverse events leading to discontinuation | 1 | 1 | 0 | 1 | 0

18. Secondary Outcome: The Percentage of Subjects With Adverse Events (AEs), Serious Adverse Events (SAEs), and AEs Leading to Discontinuation
Description: as for outcome 17
Time Frame: Up to Week 5
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | SUN-101 Via eFlow Nebulizer | SUN-101 Via eFlow Nebulizer With Activated Charcoal | Seebri® Breezhaler® | Seebri® Breezhaler® With Activated Charcoal | : Glycopyrrolate Injection
Number analyzed (Participants) | 29 | 29 | 28 | 27 | 27
percentage of participants
  Adverse Events | 20.7 | 31.0 | 25.0 | 40.7 | 25.9
  Serious Adverse Events | 0 | 0 | 0 | 0 | 0
  Adverse events leading to discontinuation | 3.4 | 3.4 | 0 | 3.7 | 0

ADVERSE EVENTS:
Time Frame: up to week 5
Description: A serious adverse event (SAE) is any SAE that occurred on or after the first dose of study medication, any SAE with a missing start date and a stop date on or after the first dose of study medication, or any SAE with both a missing start and stop date.
Arm/Group | SUN-101 Via eFlow Nebulizer | SUN-101 Via eFlow Nebulizer With Activated Charcoal | Seebri® Breezhaler® | Seebri® Breezhaler® With Activated Charcoal | : Glycopyrrolate Injection
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29 | 0/28 | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 1/29 | 3/29 | 3/28 | 5/27 | 4/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SUN-101 Via eFlow Nebulizer (N=29) | SUN-101 Via eFlow Nebulizer With Activated Charcoal (N=29) | Seebri® Breezhaler® (N=28) | Seebri® Breezhaler® With Activated Charcoal (N=27) | : Glycopyrrolate Injection (N=27)
back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
headache (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1) | 4 (4) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish.